CLINICAL TRIAL: NCT06721572
Title: Role of Home-Based Transcutaneous Electrical Acustimulation for Treatment of Pain in Patients With Chronic Pancreatitis (TEA-CuP): A Double-Blind, Sham-Controlled Crossover Trial
Brief Title: Role of Home-Based Transcutaneous Electrical Acustimulation for Treatment of Pain in Subjects With Chronic Pancreatitis
Acronym: TEA-CuP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Jorge Machicado, MD, MPH, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00260188; 025780 (Other: American College of Gastroenterology)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pancreatitis; Pancreatitis
Keywords: Abdominal Pain; Transcutaneous Electrical Acustimulation; Acupuncture; Chronic Pain
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Abdominal Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1 allocation ratio to one of two treatment sequences: i) active-TEA in treatment period 1 (week 1-4), followed by sham-TEA in treatment period 2 (week 7-10), or ii) sham-TEA in treatment period 1 (week 1-4), followed by active-TEA in treatment period 2 (week 7-10).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will receive sham or active TEA with an identical device and set of electrodes. Outcomes will be assessed via self-reported surveys. The study coordinator will be unblinded to the randomized treatment assignment. The study coordinator will implement the randomization, conduct the active and sham TEA instruction sessions, and answer study-related questions to patients. The study coordinator will not be involved in the data analysis and will not reveal treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active TEA first followed by sham TEA (Experimental): Subjects will undergo active TEA for 4 weeks (week 1-4) followed by a 2-week washout period and then sham TEA for 4 weeks (week 7-10). Subjects will have two instruction visits, one before starting active TEA and one before starting sham TEA.
  Interventions: Device: TEA
- Sham TEA first followed by active TEA (Experimental): Subjects will undergo sham TEA for 4 weeks (week 1-4) followed by a 2-week washout period and then active TEA for 4 weeks (week 7-10). Subjects will have two instruction visits, one before starting active TEA and one before starting sham TEA.
  Interventions: Device: TEA

INTERVENTIONS:
Device: TEA — Active TEA or sham TEA will be self-administered at home over two daily treatment sessions of 30 minutes each in the morning and evening. Active TEA will be delivered through an active stimulation acupoint that has previously shown to reduce abdominal pain in other patient populations. Sham TEA will be administered at a different point a few cm away from the active site and that has been shown to be ineffective in reducing pain. Other than the location, the anatomical location, application of TEA and sham will be identical. The device will be programmed by the study team to generate fixed frequency, pulse width, and time on/time off during the pulsed stimulation. The subject is only able to change the stimulation output in a range from 0-10 milliampere.

SUMMARY:
Transcutaneous Electrical Acustimulation (TEA) is a noninvasive acupuncture method that can be self-administered at home without needles. TEA transmits a weak electrical current using electrodes placed at acupoints and has shown to safely reduce pain in other gastrointestinal conditions. This study will help elucidate if TEA is effective in treating abdominal pain in patients with painful chronic pancreatitis (CP).

DETAILED DESCRIPTION:
Pain in patients with CP is debilitating and impairs quality of life. Despite using medical, endoscopic, or surgical treatments, many patients continue experiencing substantial pain and some are prescribed long-term opioids. This clinical trial aims to assess the analgesic effect of a mild electrical stimulator called TEA. TEA consists of a small, wearable device that can be used at-home while doing daily activities. If effective, this could be an alternative non-pharmacological and non-invasive option to manage pain related to CP.

In this study, the investigators will conduct a randomized, sham-controlled, 2x2 crossover trial in patients with painful CP. Subjects will be randomized to receive either active TEA first followed by sham TEA, or sham TEA first followed by active TEA. Other than the application point in the skin, active and sham TEA will be identical. The study will examine the effect of TEA on pain severity (primary outcome), pain interference and overall pain experience (secondary outcomes). The study will be conducted over 12 weeks in 5 periods: run-in (1 week), treatment period 1 (4 weeks), washout (2 weeks), treatment period 2 (4 weeks), and close-out visit (1 week). Subjects will complete online questionnaires about pain and health throughout the duration of the study. There will be a total of 3 study visits that will be conducted at the main Ann Arbor Hospital or virtually. All the study tasks can be completed remotely. The study will recruit patients from a single clinical center and from self-referral from patients with CP in the US. The proposed study will advance our understanding on the role of TEA for non-opioid pain management of CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or suspected Chronic Pancreatitis (CP). Definite CP features include presence of pancreatic calcifications or Cambridge grade 3-4 on imaging. Suspected CP features include presence of Rosemont criteria suggestive of CP on endoscopic ultrasound or 2 documented attacks of acute pancreatitis separated by at least 1 month without other definite or suspected CP features.
* Abdominal pain that is present for at least 3 months prior to enrollment and having experienced moderate intensity abdominal pain (rated as 4 or higher on a 0-10 Numeric Rating Scale) at least once in the last month.

Exclusion Criteria:

* Breastfeeding mother
* Pregnant or intending to become pregnant within the next 3 months
* Incarcerated individuals
* Unwillingness or inability to consent
* Unable to read and speak English precluding completion of questionnaires.
* Familiarity with acupoints that limit blinding
* Currently receiving acupuncture therapy
* Participation in another clinical trial
* Undergoing treatment for cancer or has a suspected or confirmed diagnosis of pancreatic cancer
* Substantial cognitive impairment or mental illness that would prevent providing informed consent and completion of questionnaires.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study
* History of total pancreatectomy with or without islet autotransplantation
* Had during the past month or plan to have within the next 3 months at least one of the following procedures: endoscopic retrograde cholangiopancreatography, pancreatic pseudocyst drainage, celiac plexus block or neurolysis, extracorporeal shock wave lithotripsy, or surgical pancreatic resection or drainage procedure
* Presence of obstructed pancreatic duct that has not yet undergone an attempt for ductal decompression.
* Known allergy to adhesive Electrocardiogram (ECG) electrodes
* History of vagal nerve surgery
* History of bilateral below the knee amputation
* History of lower extremity paralysis
* Presence of an implantable electrical stimulation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Difference of the difference of the Pain Severity Score based the Brief Pain Inventory-Short Form (BPI-SF) between start and end of each treatment period | Baseline-4 weeks and weeks 6-10
  The 4 pain intensity items (worst, least, average, and current pain) are rated on an 11-point numerical rating scale (0 = no pain, 10 = worst possible pain). A Pain Severity Score is calculated by adding the scores for the 4 items pertaining to pain intensity and then dividing this by 4. A higher number indicates higher levels of pain.

SECONDARY OUTCOMES:
Difference of the difference of the Pain Interference Score on BPI-SF between start and end of each treatment period | Baseline-4 weeks and weeks 6-10
  The BPI-SF pain interference subscale includes 7 items evaluating the impact of pain on sleep, mood, walking ability, general activity, work, relationships, and enjoyment of life over the past 1 week rated on an 11-point scale from 0 = does not interfere to 10 = completely interferes. A Pain Interference Score is calculated by adding the scores for the 7 items pertaining to pain interference and then dividing by 7. This gives an interference score from 0 to 10 (higher score indicating more interference)
Difference of the difference of the average worst daily abdominal pain using a numeric rating scale (0-10) between start and end of each treatment period (baseline-4 weeks and weeks 6-10) | Baseline-4 weeks and weeks 6-10
  This will be based on using a numeric rating scale (0-10) with higher scores indicating more pain.
Difference of the difference of the Change of Comprehensive Pain Assessment Tool Short Form (COMPAT-SF) score between start and end of each treatment period | Baseline-4 weeks and weeks 6-10
  The COMPAT-SF carries 5 sub-scores for pain pattern, pain severity, pain provocation, pain spreading, and pain description, with higher scores denoting worse pain. Participants will complete 6 questions. A) The pain pattern scale ranges from 50-100; B) severity score ranges from 0-100; C) provocation score ranges from 0-70; D) spreading score ranges from 0-90 and E) description score ranges from 0-80. A total score ranges from 0-90 with higher scores denoting worse pain.
Patient Global Impression of Change (PGIC) at end of each treatment period between the intervention group and sham group | 4 weeks and 10 week
  PGIC is a 1-item survey that measures patient perceptions of intervention success. This uses a 7-point Likert scale that will be used to asses analgesic response to TEA: 1) very much improved; 2) much improved; 3) minimally improved; 4) no change; 5) minimally worse; 6) much worse; and 7) very much worse.
Predict difference of the difference of Pain Severity Score using pain widespreadedness at beginning of each treatment period | Baseline-4 weeks and weeks 6-10
  Baseline pain before each treatment period will be classified as 'localized' or 'widespread' using a body map. This will be used to predict change of pain severity score (pre minus post) assessed by BPI-SF.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge D Machicado, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No